CLINICAL TRIAL: NCT07141836
Title: Evaluation of the Effectiveness ff Elastic Chains Versus Elastics in Maxillary Canine Retraction: A Randomized Clinical Trial
Brief Title: Effectiveness of Elastic Chains Versus Elastics in Maxillary Canine Retraction
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Asraa Haleem Mohamed Tah, Resident in orthodontics, Sana'a University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Asraa-H-Ortho
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Elastic Chains; Elastics
Keywords: Elastics; Elastomeric chains; Randomized clinical trial; Split mouth; Digital models; Canine retraction
MeSH Terms: interventions — Elasticity

STUDY DESIGN:
Intervention Model Description: This study was designed as a split-mouth randomized clinical trial, where each participant received both interventions. One side of the maxillary arch was retracted with elastic chains, while the contralateral side received elastics. This design allows for direct intra-individual comparison between the two force delivery systems.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the clinical intervention, neither the patients nor the investigator could be blinded to the treatment. However, researcher blinding was implemented at the data measurement stage through coding of OPG images and dental models by inter examiner, before measurements began. The researcher was blinded to patient identities and the type of retraction method used on each side (elastic chain vs. elastics).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic chains (Experimental): This side received maxillary canine retraction using elastic chains
  Interventions: Procedure: Elastomeric chain
- Elastics (Experimental): This side received maxillary canine retraction with Elastics on the contralateral side of the arch
  Interventions: Procedure: Elastics

INTERVENTIONS:
Procedure: Elastomeric chain — Elastic chain used to apply force that is capable of canine retraction. The chains were attached between canine bracket and molar band on the side that selected Randomly.
  Other Names: Elastic chains; Power chain
  Arms: Elastic chains
Procedure: Elastics — Elastics were used to bring a continuous force for maxillary canine retraction in orthodontic patients. Elastics were stretched between the canine bracket and the molar band to retract the canine distally
  Other Names: Elastic band; Intramaxillary elastic
  Arms: Elastics

SUMMARY:
This clinical study aimed to evaluate the effectiveness of Elastics and Elastic chains in maxillary canine retraction. Participants of this study were patients undergoing maxillary canine retraction after first premolar extraction. The study aimed to determine an effective method for better controlling tooth movement.

This study was initiated on 01-2024. Initially, I was not aware of the importance of early registration on ClinicalTrials.gov. Registration was completed after the study began to ensure transparency and adherence to ethical guidelines. All study procedures and protocols have been conducted under the supervision of the academic advisor. All study procedures and protocols have been followed according to institutional and ethical guidelines

DETAILED DESCRIPTION:
This split-mouth Randomized clinical trial was conducted on 33 patients who needed maxillary canine retraction. Participants were randomly selected one side to receive an elastic chain and the other for elastics, as a method for canine retraction. The intervention period lasted for 15 weeks, and the elastics were replaced by the patient every three days, while elastic chains were exchanged by the principal investigator at 5-week appointments. The type of movement that occurred with each method was evaluated to measure the rate of tooth movement, tipping, and rotation resulting. The study was conducted under the supervision and approval of the Research Ethics Committee at Sana'a University, Faculty of Dentistry. All procedures were performed according to the approved protocol, ensuring participant safety and data accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients' treatment required 1st premolar extractions in the maxillary arch and space closure involving canine retraction.
* Teeth in the buccal segments were without any gross anatomic root anomalies as determined by panoramic radiographs.
* There is no gross evidence of asymmetric bone loss in the buccal segments of a given arch as determined by panoramic radiographs.
* Crown/root ratios of contralateral canines and premolars are within 3 mm of one another as determined by panoramic radiographs.

Exclusion Criteria:

* Patients with gross anatomical anomalies in upper maxillary canines
* Patients with growth and development problems.
* Evidence of bone loss.
* Presence of Impacted Canine.
* History of long-term use of NSAIDs and corticosteroids or drugs affect bone metabolism. Patients who reported any medication interfering with bone metabolism or patients with severe skeletal discrepancies indicated for orthognathic treatment.
* Patients with latex materials allergy.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of maxillary canine retraction by elastics and elastic chains on each side | Difference between pe and post retraction canine position during 15 weeks
  The canine retraction rate was measured on superimposed digital casts of pre and post retraction models.
Measurement of the Tipping movement occurred by each method | Pre and post retraction during 15 weeks
  Tipping angle on each side was measured on Orthopantomograms (OPG).
Measurements of rotation resulted by elastic and elastic chain | Pre and post-retraction during 25 weeks
  The rotational angle was measured on each side by the digital models

CONTACTS AND LOCATIONS:
Overall Officials: Asraa H Taha, MSc Student, Principal Investigator — Faculty of Dentistry - Sana'a University; Reema A Al-Eriani, PhD of Pedodontics, Study Director — Faculty of Dentistry- Sana'a University; Ghamdan A Al-Harazi, PhD of Orthodontics, Study Director — Faculty of Dentistry- Sana'a University
Locations (1):
- Deparyment of Orthodontics - Faculty of Dentistry- Sana'a University, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Yes
I plan to share de-identified individual participant data (IPD) related to the main outcomes of this study. The data will be available upon reasonable request and after the results are published. Only researchers with valid proposals will be allowed access. Data will be shared through secure methods and only for academic purposes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: 01-Jan-2026 End Date: 31-Dec-2030
Access Criteria: Qualified researchers who submit a valid research proposal will be able to access de-identified individual participant data, including digital models and treatment outcome measurements. Data will be available through a secure online repository upon approval of the research proposal.

REFERENCES:
- [Result] Jagtap SB, Bhosale VI, Patil AS. Comparative evaluation of interrupted and intermittent forces on canine retraction: an in vivo study. Folia Med (Plovdiv). 2021 Oct 31;63(5):686-691. doi: 10.3897/folmed.63.e54247. PMID 35851202
- See also: Comparative evaluation of interrupted and intermittent forces on canine retraction: an in vivo study — https://pubmed.ncbi.nlm.nih.gov/35851202/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT07141836/Prot_ICF_000.pdf